CLINICAL TRIAL: NCT01167790
Title: Interest of Oral Tissue Autofluorescence for the Screening of Precancerous Lesions and Cancer in Population With Tobacco and Alcohol Abuse.
Brief Title: Autofluorescence for the Screening of Precancerous and Malignant Lesions
Acronym: FLUOK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2010/02
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Precancerous Lesions of the Oral Mucosa
Keywords: Precancerous lesions of the oral mucosa; Fluorescence visualization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: buccal cavity examination — autofluorescence examination

SUMMARY:
Diagnosis of oral squamous cell carcinoma is always too late. Due to this delay for diagnosis, prognosis is very bad. It has been demonstrate that systematic oral examination decrease mortality in tobacco and alcohol consumers population (Sankaranarayanan and al. Lancet 2005, 4, 1927-1933 ). An other study has demonstrate that autofluorescence is a useful technic for detection of dysplasia and squamous cell carcinoma that cannot be seen with conventional oral examination((Poh CF Wink Cancer Res on 2006 ( 22 ): 6616-22; Poh CF Head Neck 2007 ( 1 ) 7 71-6).However autofluorescence has never been evaluated has a screening tool for systematic oral examination and the reproductibility has never been studied.

DETAILED DESCRIPTION:
The study of Sankaranarayanan and al. (Lancet on 2005, 4, 1927-1933) demonstrated the influence on the decline of mortality of a realized systematic screening, by a simple visual inspection of the oral cavity in alcohol-smoker patients. The sensibility of the visual inspection to diagnose the oral cancers is estimated at 85 % and the specificity in 97 %. However some lésions are not diagnosed with common oral examination(Downer MC Oral Oncol. 2004 ( 3 ) 264-73). The examination in autofluorescence coupled with the visual inspection could be a solution to improve early diagnosis of potentially malignant disorders . Indeed, dysplasia and cancerous lesions can be revealing by an autofluorescence examination (Lane PM J Biomed opt on 2006 ( 2 ): 024006). Other works demonstrated that infra-clinical lesions could be revealed by the autofluorescence (Poh CF Wink Cancer Res on 2006 ( 22 ): 6616-22; Poh CF Head Neck 2007 ( 1 ) 7 71-6). On the other hand the sensibility and the specificity of the autofluorescence in situation of screening were not estimated and studies carried out on sick subjects tend to overestimate the metrological performances of a technique. Besides the reliability of the technique (reproducibility) was not studied. For these reasons, it is recommended to realize in situation of screening in an alcohol-smoker population:

* a study of reliability to estimate the reproducibility inter-observer of the examination of the oral cavity in tissular autofluorescence and,
* a feasibility study to estimate the potential contribution of the autofluorescence with regard to a simple visual inspection in the screening of the potential malignant disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized for alcoholic weaning
* consumption activates of tobacco or stop for less than one year
* consent form signed

Exclusion Criteria:

* patient presenting a disorder of the haemostasis (plaques < 50G / L; INR > 3, haemophilia, moderate or severe Willebrand disease),
* absorption of acid acetylsalicylic in seven days before inclusion,
* the patient with oral cavity precancerous pathology, dysplasia or known cancer patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
reliability | one day
  Concordance inter-observer, considered by the coefficient kappa of Cohen, towards the decision to make a biopsy of a suspicious lesion(potentially malignant lesions, dysplasia and cancer)

SECONDARY OUTCOMES:
Prevalence | one day
  Prevalence of potentially malignant lesions, dysplasia and cancer patient of the oral cavity in conditions of screening in an alcoolo-smoking population.
Validity | one day
  anatomopathologic diagnosis wil be compared to examination in both techniques of examination
safety | one day
  adverse events of the procedure (biopsy)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-chritophe FRICAIN, Md-PhD, Principal Investigator — University Hospital, Bordeaux; Adélaïde DOUSSAU, MD, Study Chair — University Hospital, Bordeaux; Jean-christophe FRICAIN, MD-PhD, Study Director — University Hospital, Bordeaux
Locations (1):
- Hopital Saint André, Bordeaux, France